CLINICAL TRIAL: NCT03783767
Title: Peer Leadership for Physical Literacy: A Randomized Controlled Trial for Elementary School Students
Brief Title: Peer Leadership for Physical Literacy
Acronym: PLPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other); University of Victoria (Other); Newcastle University (Other)
Responsible Party: Principal Investigator, Mark Beauchamp, Professor of Kinesiology, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H18-00141
Record Dates: First submitted 2018-12-17; First posted 2018-12-21 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Leadership; Physical Activity
Keywords: school; intervention; physical literacy; peer mentor; leadership; motor skills; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leadership Intervention Group (Experimental): Teachers in the intervention group will receive a half day workshop from a member of the research team. These teachers will then provide a four week training program to Grade 6/7 students, who will then deliver a 10-week fundamental movement skill (FMS) training program to Grade 3/4 students.
  Interventions: Behavioral: Leadership Intervention
- Waitlist Control (No Intervention): This group of students and teachers will act as a waitlist control group. Therefore, during the same time that the other group is receiving the intervention, this group will proceed with their normal practices.

INTERVENTIONS:
Behavioral: Leadership Intervention — Grade 6/7 teachers will take part in a workshop on developing transformational leadership among their Grade 6/7 students, and provide teachers with a 4-week training program. Teachers will implement a 4-week leadership development component to their Grade 6/7 students. Grade 6/7 students will then deliver a 10-week peer-led FMS program to Grade 3/4 students. The Grade 6/7 peer leaders will lead 2 x 30 min sessions per week during physical education classes, recess, or lunch times. In weeks two and three, peer leaders will be observed by members of the research team and provided with feedback using a structured checklist regarding their delivery in the session. Mid-way through the 10-week program teachers will deliver a booster leadership training component to the Grade 6/7 peer-leaders.
  Arms: Leadership Intervention Group

SUMMARY:
The purpose of the proposed research is to develop, implement, and test the efficacy of a theory-driven evidence-based peer leadership program for elementary school students (Grade 6/7; age 11/12 years) in relation to (a) their own leadership skills and their leadership self-efficacy (i.e., confidence to lead), as well as (b) the physical literacy of younger (Grade 3/4; age 8/9) students with whom they are partnered.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be teachers (Grade 6/7) and students (Grade 3,4, 6 or 7) in elementary schools in the Lower Mainland of British Columbia.
* Students must have a basic working knowledge of English.

Exclusion Criteria:

* There are no exclusion criteria that would exclude anyone who otherwise meets the inclusion criteria specified above

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 359 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Teacher's rating of their student's transformational leadership using the Transformational Teaching Questionnaire | Change from Baseline Transformational Leadership at 6 months (Post Intervention)
  Transformational leadership by Grade 6/7 peer leaders will be assessed by teachers using an adaption version of the Transformational Teaching Questionnaire (Beauchamp et al., 2010). This abbreviated measures has been used in our previous studies which demonstrated sound reliability (cronbach alpha > 0.89).

SECONDARY OUTCOMES:
Self-Rated Leadership Self-Efficacy using a ten-item questionnaire | Change from Baseline Leadership Self-Efficacy at 6 months (Post Intervention)
  Leadership Self-Efficacy by Grade 6/7 peer leaders will be assessed using a ten-item leadership self-efficacy measure using Bandura's (2006) recommended procedures for assessing self-efficacy.
Grade 3/4 student self reported intrinsic motivation using the Intrinsic motivation measure by Sebire and colleagues (2013) | Change from Baseline Intrinsic Motivation at 6 months (Post Intervention)
  Intrinsic motivation among Grade 3/4 students will be assessed using the Intrinsic Motivation measure developed by Sebire and colleagues (2013) for specific use with young children in school physical education settings. This measure displays sound reliability (cronbach alpha = 0.77), as well as factorial validity.
Grade 3/4 self-reported Perceived Competence using the Perceived Competence measure developed by Sebire and colleagues (2013) | Change from Baseline Intrinsic Motivation at 6 months (Post Intervention)
  Grade 3/4 Perceived Competence will be measured by a questionnaire developed by Sebire and colleagues (2013) for specific use in school physical education settings with young children. This measure has been shown to display sound reliability (cronbach alpha = 0.72).
Physical Self Description Questionnaire (Marsh et al., 2010) will assess Grade 3/4 self-reported self-concept | Change from Baseline Self-Concept at 6 months (Post Intervention)
  The Physical Self Description Questionnaire is a self-report measure for Grade 3/4 students that has sound reliability and factorial validity.
Fundamental Movement Skills Competence assessed via the Test of Gross Motor Development (3rd edition) and product scores (throw/kick speed, successful number of catches) | Change from Baseline Fundamental Movement Skills at 6 months (Post Intervention)
  The kick, throw and a combination throwing/catching test will be performed. Skills will be videoed so that raters can assess the process of each movement and score according to predefined criteria of the Test of Gross Motor Development 3rd edition (Ulrich and Webster, 2017). Our assessment will also enable us to assess maximal kicking and throwing speed. The combination throwing/catching test will be performed for two trials of 30 seconds each, with scores assigned based on the number of successful catches each participant completes.
School Day Physical Activity will be assessed in Grade 3/4 students using hip worn GT3X+ accelerometers | Change from Baseline School Day Physical Activity at 6 Months (Post Intervention)
  A subsample of Grade 3/4 students will be randomly selected to wear an accelerometer for one school week (5 days) during the school day only.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Beauchamp, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Psychology of Exercise, Health, and Physical Activity Laboratory, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nathan N, Sutherland R, Beauchamp MR, Cohen K, Hulteen RM, Babic M, Wolfenden L, Lubans DR. Feasibility and efficacy of the Great Leaders Active StudentS (GLASS) program on children's physical activity and object control skill competency: A non-randomised trial. J Sci Med Sport. 2017 Dec;20(12):1081-1086. doi: 10.1016/j.jsams.2017.04.016. Epub 2017 Apr 21. PMID 28487140
- [Background] Beauchamp MR, Barling J, Li Z, Morton KL, Keith SE, Zumbo BD. Development and psychometric properties of the transformational teaching questionnaire. J Health Psychol. 2010 Nov;15(8):1123-34. doi: 10.1177/1359105310364175. Epub 2010 Jun 3. PMID 20522503
- [Background] Sebire SJ, Jago R, Fox KR, Edwards MJ, Thompson JL. Testing a self-determination theory model of children's physical activity motivation: a cross-sectional study. Int J Behav Nutr Phys Act. 2013 Sep 26;10:111. doi: 10.1186/1479-5868-10-111. PMID 24067078
- [Background] Marsh HW, Martin AJ, Jackson S. Introducing a short version of the physical self description questionnaire: new strategies, short-form evaluative criteria, and applications of factor analyses. J Sport Exerc Psychol. 2010 Aug;32(4):438-82. doi: 10.1123/jsep.32.4.438. PMID 20733208
- [Derived] Hulteen RM, Lubans DR, Rhodes RE, Faulkner G, Liu Y, Naylor PJ, Nathan N, Waldhauser KJ, Wierts CM, Beauchamp MR. Evaluation of the peer leadership for physical literacy intervention: A cluster randomized controlled trial. PLoS One. 2023 Feb 16;18(2):e0280261. doi: 10.1371/journal.pone.0280261. eCollection 2023. PMID 36795739

DOCUMENTS (1):
  • Study Protocol (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT03783767/Prot_000.pdf